CLINICAL TRIAL: NCT00136643
Title: A Phase I/II Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Tolerance and Acceptability of a Vaginal Gel Containing Sodium Lauryl Sulfate (Invisible Condom®) in Healthy Female Subjects
Brief Title: Safety, Tolerance and Acceptability Trial of the Invisible Condom® in Healthy Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Centre Hospitalier de l'Universite Laval (CHUL) (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CRI-INV.06; FRN: 67531
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: microbicide; Women; Prevention; HIV; STIs; HIV Seronegativity; prevention of sexually transmitted infections including HIV.
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

INTERVENTIONS:
Drug: Invisible Condom®

SUMMARY:
The objectives of this clinical study are to evaluate the extended safety, tolerance and acceptability of a vaginal gel formulation when applied in 452 healthy women volunteers. This vaginal formulation was shown to be well tolerated in a previous smaller clinical study. The formulation is being developed as a microbicide for the prevention of sexually transmitted infections (STIs) including HIV.

DETAILED DESCRIPTION:
Objectives: The objectives of this Phase I/II clinical trial are to evaluate the safety, tolerance and acceptability of a gel formulation containing sodium lauryl sulfate (SLS) (compared to gel alone and placebo) when applied intravaginally in healthy volunteers.

Design: In part A of the protocol, three groups: gel alone, gel plus SLS, and placebo will be tested for safety, tolerance and acceptability when applied intravaginally once, twice or three times daily for 14 days in 252 healthy subjects. The volunteers will be divided as follow: 36 sexually abstinent healthy subjects (12 per group) will apply the gel, gel plus SLS or the placebo once daily for 14 days; 72 sexually active healthy subjects (24 per group) will apply the gel, gel plus SLS or the placebo once daily for 14 days; 72 sexually active healthy subjects (24 per group) will apply the gel, gel plus SLS or the placebo twice daily for 14 days and 72 sexually active healthy subjects (24 per group) will apply the gel, gel plus SLS or the placebo three times daily for 14 days. The gel will be applied between menses. For the sexually active group, the gel should be applied less than 1 hour before sexual intercourse, if planned. Subjects will have vaginal intercourse a minimum of 4 times in a 2-week period of gel application.

In part B of the protocol, the extended safety of the gel alone, gel plus SLS and placebo will be studied when applied intravaginally twice daily for 8 weeks in sexually active healthy subjects. In this part B (actually represents Phase II of the trial), 80 healthy sexually active subjects for the gel alone group and 80 subjects for the gel + SLS group and 40 subjects for the placebo group, will be studied. The part B involves the participation of a total of 200 subjects. Subjects will have vaginal intercourse a minimum of 4 times in a 2-week period of gel application. The gel will be applied between menses. The gel should be applied less than 1 hour before sexual intercourse, if planned, but no more than twice a day.

ELIGIBILITY:
Inclusion Criteria:

* Sign an informed consent
* Healthy female subjects aged between 18 to 49. Healthy female subjects are defined as individuals who are free from clinically significant illness or disease as determined by their medical history, physical examination and laboratory tests.
* Normal physical and gynecological examinations
* Normal colposcopic examination
* Have regular menstrual cycle with 21-40 days between menses
* HIV-negative subjects and at low risk of acquiring HIV
* At low risk of getting STIs (i.e. sexually abstinent or having history of protected sexual intercourse or having a stable sexual partner). Sexual intercourse is defined here as vaginal penetration. Stable sexual partner is defined as the same sexual partner for the length of the study.
* Agreeing to abstain from sexual intercourse from screening to the end of the study (for sexually abstinent subjects).
* Agreeing to have sexual intercourse a minimum of 4 times for each period of two weeks of gel application (for sexually active subjects)

Exclusion Criteria:

* Clinically significant abnormal physical and/or gynecological examination
* Clinically significant abnormal laboratory findings
* Allergy to applicator material (polyethylene) or to gel polymer (polyoxyethylene-polyoxypropylene) or to latex
* Participation in any investigational study involving drugs, vaccines or microbicides in the last 30 days
* History of toxic shock syndrome
* HIV infection
* Bacterial vaginosis or Candida or Trichomonas vaginitis at time of screening
* STIs (gonorrhea, chlamydia, syphilis, genital herpes, chancroid) at time of screening
* Breakthrough menstrual bleeding, or vaginal bleeding during or following sexual intercourse, in the last 3 months
* Intravenous (IV) drug use except for medical reasons in the last year
* Pregnant at enrolment or breast-feeding
* Having received antibiotics in the last 14 days
* Subjects considered as unreliable or unable to understand or follow the study protocol directions
* Use of an intrauterine device

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 452
Dates: Start 2005-06; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerance outcomes: Subjective assessment; Objective assessment

SECONDARY OUTCOMES:
Acceptability assessment

CONTACTS AND LOCATIONS:
Overall Officials: Michel G. Bergeron, MD, FRCPC, Principal Investigator — Prof. and Director of Infectious Diseases Research Center, Laval University
Locations (1):
- Laboratoire de Santé Hygiène Mobile, Yaoundé, Cameroon